CLINICAL TRIAL: NCT02804867
Title: A Blood Test to Identify Persons at Risk of Developing Depression or Bipolar Disorder
Brief Title: Spot Depression Study
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Jordan Ramsey, Postdoctoral researcher, University of Cambridge
Other Study IDs: HBREC.2015.06
Record Dates: First submitted 2016-06-07; First posted 2016-06-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder; Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Depression
  Interventions: Procedure: Online questionnaire and self-administered blood spot
- Bipolar disorder
  Interventions: Procedure: Online questionnaire and self-administered blood spot
- Control
  Interventions: Procedure: Online questionnaire and self-administered blood spot

INTERVENTIONS:
Procedure: Online questionnaire and self-administered blood spot

SUMMARY:
This study aims to identify signs of depression and bipolar disorder by measuring changes of certain molecules (biomarkers) that can be detected in dried blood spots. Our goal is to use these biomarkers to develop a diagnostic test to enable early treatment, which can lead to better patient outcomes.

DETAILED DESCRIPTION:
Bipolar disorder and major depression are serious mental health conditions that have a devastating impact on patients, their families and friends, and society. Currently, no laboratory test exists for these disorders. We are trying to develop a molecular test based on blood spots (small spots of blood obtained from patients' fingertips that have been dried on special paper). Volunteers take part by filling out the questionnaire at www.spot-depression.org. They may then be selected to provide a dried blood spot, which can be collected at home using a kit that will be mailed to their address.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the United Kingdom
* Over 18 years of age

Exclusion Criteria:

* Pregnant or breastfeeding
* Presence of blood-borne infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited using flyers, emails, and online recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Comparison of protein concentrations in dried blood spots between patient groups and controls | Baseline (at enrollment); no follow-up
Assessment of classification accuracy of protein concentrations in dried blood spots for distinguishing between bipolar disorder and depression | Baseline (at enrollment); no follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Bahn, MD/PhD, Principal Investigator — Principal Investigator
Locations (1):
- Jordan Ramsey, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No